CLINICAL TRIAL: NCT04968184
Title: A Phase 3 Randomized Double-Blind Placebo-Controlled Multicenter Study to Assess the Efficacy and Safety of KBP-5074 Mineralocorticoid Receptor Antagonist in Subjects With Uncontrolled Hypertension and Moderate or Severe (Stage 3b/4) CKD
Brief Title: Efficacy and Safety of KBP-5074 in Uncontrolled Hypertension and Moderate or Severe Chronic Kidney Disease (CKD)
Acronym: Clarion-CKD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim futility analysis showed primary endpoint not achieved
Sponsor: KBP Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KBP5074-3-001
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Stage 3b/4 chronic kidney disease; Hypertension; Uncontrolled Hypertension; Blood pressure; Mineralocorticoid Receptor Antagonist; Randomized withdrawal
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — KBP-5074

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals directly involved in the conduct of the study, including participants, Investigators, site staff, clinical research organization (CRO) personnel, and Sponsor study personnel, will remain blinded to treatment assignments until all participants have completed the Week 56 end of study (EOS) Visit (Visit 17) and the database locked in preparation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Open-label Placebo Run-In Period: All eligible participants will receive matching placebo, for approximately 2 weeks, during the Open-label placebo Run-In period.
  Double-blind Treatment Period: All eligible participants will receive matching placebo, from week 2 thru week 24 during the Double-blind treatment Period
  Open-label Treatment Period: All eligible participants will receive KBP-5074, from week 24 thru week 48 during the Open label Treatment Period
  Randomized Double-blind Withdrawal Period: All eligible participants will be randomized to either continue their current KBP-5074 dose at the end of the Open-Label Treatment Period or receive matching placebo from week 48 thru week 52.
  Follow up Period: All participants will discontinue matching placebo/KBP-5074 and be followed for safety until end of study visit from week 52 to week 56.
  Interventions: Drug: Placebo
- KBP-5074 (Experimental): Open-label Placebo Run-In period: All eligible participants will receive matching placebo, for approximately 2 weeks during the Open-label placebo Run-In period.
  Double-blind Treatment Period: All eligible participants will receive KBP-5074, from week 2 thru week 24 during the Double-blind Treatment Period
  Open-label Treatment Period: All eligible participants will receive KBP-5074, from week 24 thru week 48 during the Open label Treatment Period
  Randomized Double-blind Withdrawal Period: All eligible participants will be randomized to either continue their current KBP-5074 dose at the end of the Open-Label Treatment Period or receive matching placebo from week 48 thru week 52.
  Follow up Period: All participants will discontinue matching placebo/KBP-5074 and be followed for safety until end of study visit from week 52 to week 56.
  Interventions: Drug: KBP-5074

INTERVENTIONS:
Drug: Placebo — Participants will orally receive placebo matching to KBP-5074 tablets QD.
  Arms: Placebo
Drug: KBP-5074 — Participants will orally receive KBP-5074 tablets, from 0.25 mg to a maximum dose of 0.5-mg QD.
  Arms: KBP-5074

SUMMARY:
This Phase 3, randomized, Double-blind, placebo-controlled, 2-arm, parallel-group, multicenter study with randomized withdrawal will evaluate the efficacy, safety, and durability of KBP-5074 in adult participants who have stage 3b/4 chronic kidney disease (CKD) (estimated glomerular filtration rate [eGFR] calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula [eGFR {EPI}] ≥15 to ≤44 mL/min/1.73 m^2) and uncontrolled hypertension (systolic blood pressure (SBP) ≥140 and <180 mm Hg and taking 2 or more antihypertensive medications.

DETAILED DESCRIPTION:
Participants in this study will be recruited, screened, and enrolled at approximately 140 study sites globally.

The study will consist of the following periods:

1. Pretreatment Phase: This will include prescreening assessment and screening period of up to 4 weeks and 2-week Open-label placebo Run-In period.
2. A 24-week Double-blind Treatment Period (Randomization to Week 24) will include: An initial 12-week (Randomization to Week 12) and second 12-week (Week 12 to Week 24) treatment period and a second 12-week treatment period (Week 12 to Week 24), during both the periods study drug will be titrated.
3. A 24-week Open-label Treatment Period (Week 24 to Week 48) during which eligible participants will receive Open-label KBP-5074.
4. A 4-week Randomized Double-blind Withdrawal Period (Week 48 to Week 52) during which eligible participants will be randomized to continue their current KBP-5074 dose at the end of Open-label treatment or receive matching placebo for 4 weeks.
5. A 4-week post-treatment Follow-Up Period (Week 52 to Week 56).

During, 24-week Double-blind Treatment Period, 24-week Open-label Treatment Period, and at 4-week Randomized Double-blind Withdrawal Period, the background antihypertensive medications change may or may not be allowed.

At Double-blind Treatment Period, eligible participants will be randomly assigned in a 1:1 ratio to KBP-5074 0.25 mg or matching placebo once daily (QD).

At the Randomized Double-blind Withdrawal Period, participants who meet the randomized withdrawal criteria will be randomly assigned in a 1:1 ratio to continue their current KBP-5074 dose at the end of the Open-label Treatment Period or matching placebo QD.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) must be ≥19 to <45 kg/m^2 at the Screening Visit
* Participant must have uncontrolled hypertension defined as meeting both of the following criteria:

  * The participant has a resting seated trough cuff SBP ≥140 mm Hg at the Screening Visit (Visit 1), and at the start (Visit 2) and end (Visit 3) of the Run-In Period
  * The participant is taking 2 or more antihypertensive medications that have been titrated upward as tolerated to hypertension target doses per local SoC and have been stable (i.e., without any dose adjustments) from 4 weeks before the Screening Visit (Visit 1) through the end of the Run-In Period (Visit 3)
* The participant must have Stage 3b (eGFR [EPI] ≥30 and ≤44 mL/min/1.73 m^2) or Stage 4 (eGFR [EPI] ≥15 and <30 mL/min/1.73 m^2) CKD.

Exclusion Criteria:

* Participant has a resting seated trough cuff SBP ≥180 mm Hg at the Screening Visit (Visit 1) or at the start (Visit 2) or end (Visit 3) of the Run-In Period
* Participant has a serum potassium level >4.8 mmol/L during the Screening or Run-In Periods
* Participant has had a serum potassium level >5.6 mmol/L within 2 weeks before the Screening Visit (Visit 1)
* Participant has been hospitalized for hyperkalemia within the 3 months before the Randomization Visit (Visit 3)
* Participant was not compliant with taking placebo during the Run-in Period or participant was not compliant with background antihypertensive medications during the Run-in Period as assessed at the Randomization Visit (Visit 3)
* Participant has taken an mineralocorticoid receptor antagonist (MRA), a potassium-sparing diuretic, or chronic potassium supplements during the 4 weeks before the Screening Visit (Visit 1)
* Participant has taken potassium binders for the treatment of hyperkalemia during the 3 months before the Screening Visit (Visit 1)
* Participant has taken a strong cytochrome P450 (CYP) CYP3A4 inducer or strong CYP3A4 inhibitor during the 7 days before the Randomization Visit (Visit 3)
* Participant has taken a prohibited traditional Chinese medication during the 28 days prior to Screening Visit (Visit 1).
* Participant was administered any other investigational product within 4 weeks or 5 half-lives (whichever is longer) prior to the Screening Visit (Visit 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 652 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Change in seated trough cuff SBP from baseline to Week 12 | From baseline to Week 12
  Efficacy of KBP-5074 in reducing SBP by assessing change in seated trough cuff SBP for KBP-5074 dose regimen compared to placebo, will be evaluated.
Change in seated trough cuff SBP from Week 48 to Week 52 | Week 48 to Week 52
  Durability of KBP-5074 in reducing SBP by assessing change in seated trough cuff SBP for the KBP-5074 dose regimen compared to placebo, will be evaluated.

SECONDARY OUTCOMES:
Change in seated trough cuff SBP from baseline to Week 24 | From baseline to Week 24
  Efficacy and durability of KBP-5074 in reducing SBP by assessing change in seated trough cuff SBP, will be evaluated.
Changes in seated trough cuff diastolic blood pressure (DBP) from baseline to Week 12 and Week 24 | From baseline to Week 12 and Week 24
  Effect of KBP-5074 on DBP by assessing change in seated trough cuff DBP, will be evaluated.
Changes in seated trough cuff SBP and DBP from baseline to Week 48 | From baseline to Week 48
  Effect of KBP-5074 on SBP and DBP by assessing change in seated trough cuff SBP and DBP, will be evaluated.
Changes in urinary albumin: creatinine ratio (UACR) from baseline to Week 12 and Week 24 for participants with UACR ≥30 mg/g at baseline | From baseline to Week 12 and Week 24
  Effect of KBP-5074 on UACR by assessing changes in UACR for participants with UACR ≥30 mg/g at baseline, will be evaluated.
Percentage changes in UACR from baseline to Week 12 and Week 24 for participants with UACR ≥30 mg/g at baseline | From baseline to Week 12 and Week 24
  Effect of KBP-5074 on UACR by assessing percentage changes in UACR for participants with UACR ≥30 mg/g at baseline, will be evaluated.
Changes in UACR from baseline to Week 12, Week 24, and Week 48 | From baseline to Week 12, Week 24, and Week 48
  Effect of KBP-5074 on UACR by assessing changes in UACR for participants with macroalbuminuria (defined as UACR ≥300 mg/g) and microalbuminuria (defined as UACR ≥30 and <300 mg/g) at baseline, will be evaluated.
Percentage changes in UACR from baseline to Week 12, Week 24, and Week 48 | From baseline to Week 12, Week 24, and Week 48
  Effect of KBP-5074 on UACR by assessing percentage changes in UACR for participants with macroalbuminuria (defined as UACR ≥300 mg/g) and microalbuminuria (defined as UACR ≥30 and <300 mg/g) at baseline, will be evaluated.
Change in seated trough cuff DBP from Week 48 to Week 52 | Week 48 to Week 52
  Effect of KBP-5074 on DBP by assessing change in seated trough cuff DBP, will be evaluated.
Change in UACR from Week 48 to Week 52 | Week 48 to Week 52
  Effect of KBP-5074 on UACR by assessing changes in UACR for participants with UACR ≥30 mg/g, macroalbuminuria (defined as UACR ≥300 mg/g) and microalbuminuria (defined as UACR ≥30 and <300 mg/g) at baseline, will be evaluated.
Percentage change in UACR from Week 48 to Week 52 | Week 48 to Week 52
  Effect of KBP-5074 on UACR by assessing percentage changes in UACR for participants with UACR ≥30 mg/g, macroalbuminuria (defined as UACR ≥300 mg/g) and microalbuminuria (defined as UACR ≥30 and <300 mg/g) at baseline, will be evaluated.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Screening (Week -6 to -2) until EOS (Week 56) or Unscheduled visit or end of treatment or early termination
  The safety and tolerability of KBP-5074,will be evaluated.

CONTACTS AND LOCATIONS:
Locations (215):
- United States (65):
  - G & L Research, LLC, Foley, Alabama
  - Apogee Clinical Research, LLC, Huntsville, Alabama
  - Aventiv Research, Inc, Mesa, Arizona
  - National Heart Institute, Beverly Hills, California
  - Amicis Research Center (Valencia), Granada Hills, California
  - Amicis Research Center, Granada Hills, California
  - Amicis Research Center, Lancaster, California
  - Renal Consultants Medical Group - Granada Hills, Northridge, California
  - United Clinical Research and Innovations, South Gate, California
  - Solano Kidney Care, Vacaville, California
  - Desert Cities Dialysis - Amethyst, Victorville, California
  - Kidney and Hypertension Center, Victorville, California
  - Davita Clinical Research-Hartford, Bloomfield, Connecticut
  - Synergy Healthcare, Bradenton, Florida
  - Homestead Associates in Research, Inc, Miami, Florida
  - Total Research Group, Miami, Florida
  - LCC Medical Research, Miami, Florida
  - Oceane 7 Medical&Research Center, Inc., Miami, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - South Florida Research Phase I-Iv, Inc., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Inpatient Research Clinic, LLC, Miami Lakes, Florida
  - New Generation Of Medical Research, Naples, Florida
  - Sarkis Clinical, Ocala, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Santos Research Center CORP, Tampa, Florida
  - Fides Clinical Research, Atlanta, Georgia
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Columbus Associates LLC, Columbus, Georgia
  - Central Georgia Kidney Specialists, Macon, Georgia
  - Clinical Investigation Specialists, Inc., Gurney, Illinois
  - Massachusetts General Hospital (MGH) - Renal Associates Clinic, Boston, Massachusetts
  - InterMed Consultants, Edina, Minnesota
  - Healthcare Research Network, Hazelwood, Missouri
  - Clinical Research Consultants, Kansas City, Missouri
  - St. Louis Heart and Vascular, P.C. (SLHV) - Christian Hospital Office, St Louis, Missouri
  - Healor Primary Care /CCT Research, Las Vegas, Nevada
  - DaVita Clinical Research (Nevada), Las Vegas, Nevada
  - NYC Health + Hospitals / Queens - Diabetes Center of Excellence, Jamaica, New York
  - Mattoo & Bhat Medical Associates, PC, Ridgewood, New York
  - Albert Einstein's College of Medicine, The Bronx, New York
  - Kidney Medical Associates, PLLC, The Bronx, New York
  - Mountain Kidney & Hypertension Associates (MKHA), P.A - Asheville, Asheville, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - Eastern Nephrology Associates - Jacksonville, Jacksonville, North Carolina
  - Eastern Nephrology Associates - New Bern, New Bern, North Carolina
  - North Carolina Nephrology P.A., Raleigh, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Gamma Clinical Research Institute, Austin, Texas
  - Davita Clinical Research El Paso, El Paso, Texas
  - Kidney Consultants of El Paso, P.A., El Paso, Texas
  - DaVita Clinical Research Houston, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Urology San Antonio - North Central, San Antonio, Texas
  - DaVita Clinical Research, San Antonio, Texas
  - Kidney Specialists of North Houston, PLLC, The Woodlands, Texas
  - Davita Norfolk Square, Norfolk, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Clinical Investigation Specialists, Kenosha, Wisconsin
  - Milwaukee Nephrologists, SC (Rich), Wauwatosa, Wisconsin
- Australia (3):
  - Renal Research, Gosford, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Heidelberg, Victoria
- Bosnia and Herzegovina (6):
  - Clinical Center University of Sarajevo, Sarajevo, Kanton Sarajevo
  - Univerzitetski klinicki centar Republike Srpske - Internal Medicine, Nephrology, Banja Luka, Republika Srpska
  - The University Hospital Foca, Foča, Republika Srpska
  - General Hospital Gradiska, Gradiška, Republika Srpska
  - General hospital Trebinje - Gastroenterology, Trebinje, Republika Srpska
  - General Hospital Tesanj, Tešanj, Zeničko-dobojski Kanton
- Bulgaria (13):
  - 5 th MHAT, Sofia, Sofia-Grad
  - Medical Center Excelsior, Sofia, Sofia-Grad
  - UMHAT St. Ekaterina, Sofia, Sofia-Grad
  - Comac Medical Ltd, Sofia, Sofia-Grad
  - Mhat Dr.Tota Venkova, Gabrovo
  - Medical Center Hera EOOD, Montana
  - UMHAT Kaspela, Plovdiv
  - Medical Center "Teodora", Rousse
  - DCC 22 - Sofia, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center ''Synexus Sofia'' EOOD, Sofia
  - University Hospital of Active Treatment Prof. Stoyan Kirkovich, Stara Zagora
  - MHAT"Sv.Anna-Varna"AD, Varna
- Canada (2):
  - Dr. Stephen S. Chow Medicine Professional Corporation, Toronto, Ontario
  - Clinical Research Solutions Incorporated, Waterloo, Ontario
- China (35):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing An Zhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital - Nephrology, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region- Nephrology, Nanning, Guangxi
  - The Affliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University (East Compus), Zhengzhou, Henan
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital/ The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Baotou Medical College, Inner Mongolia University of Science and Technology, Baotou, Nei Mongol (mn)
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Yantai Yuhuangding Hospital(Base Cpmpus), Yantai, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Sichuan Academy of Medical Sciences, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Jinhua Central Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Southwest Hospital of AMU, Chongqing
  - Shanghai Sixth People's Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
- Croatia (3):
  - University Hospital Centre Zagreb, Zagreb, City of Zagreb
  - Opca bolnica Vinkovci, Vinkovci, Osjecko-baranjska Županija
  - University Hospital Center Split, Split
- Czechia (4):
  - Nefrologie s.r.o., Prague, Praha 4
  - Nemocnice Trebic, p.o., Třebíč, Třebíč
  - IKEM, Prague
  - Alaron s.r.o., Prague
- Georgia (12):
  - LTD "High technology hospital MEDCENTER", Batumi, Adjara
  - Ltd Marnecor, Marneuli, Kvemo Kartli
  - Ministry of Defence of Georgia LEPL Giorgi Abramishvili Military Hospital, Gori, Shida Kartli
  - JSC "Evex Hospitals', Batumi
  - Aleksandre Aladashvili Clinic LLC, Tbilisi
  - LTD Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - "Pineo Medical Ecosystem"LTD, Tbilisi
  - JSC German Clinic, Tbilisi
  - National Center of Urology Named after Laur Managadze, Tbilisi
  - Bokhua Memorial Cardiovascular Centre, Tbilisi
  - Emergency Cardiology Center named by acad. G. Chapidze, Tbilisi
  - J.S.C."K.Eristavi National Center of Experimental and Clinical Surgery", Tbilisi
- Germany (8):
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen, Baden-Wurttemberg
  - Diabeteszentrum DO, Dortmund, North Rhine-Westphalia
  - DaVita Clinical Research Germany GmbH, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Mainz, Mainz, Rhineland-Palatinate
  - Charité- Universitätsmedizin Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
- Hong Kong (2):
  - Queen Mary Hospital - Medicine, Hong Kong
  - Tung Wah Hospital, Hong Kong
- Hungary (10):
  - Coromed-Smo Kft., Pécs, Baranya
  - IPR Hungary Kft., Miskolc, Borsod-Abauj Zemplen county
  - Sonocor Egészségügyi Szolgáltató Kft., Szeged, Csongrád megye
  - TaNa Med Kft, Mosonmagyaróvár, Győr-Moson-Sopron
  - BKS Research, Hatvan, Heves County
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa Hungary, Pest County
  - DRC Gyógyszervizsgáló Központ Kft., Balatonfüred, Veszprém City
  - Semmelweis Egyetem, Budapest
  - Jahn Ferenc Dél-Pesti Kórház és Rendelőintézet, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
- Israel (2):
  - Rabin Medical Center, Petah Tikwa, Central District
  - Nazareth Hospital EMMS, Nazareth, Northern District
- Latvia (2):
  - Dace Teterovska - Doctor's Practice, Ogre, Ogre
  - P.Stradina Clinical University Hospital, Riga
- Saules seimos medicinos centras, Kaunas, Kaunas County, Lithuania
- Malaysia (5):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Seri Manjung, Seri Manjung, Perak
- Poland (9):
  - NZOZ Euromedica Sp. z o.o., Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Prywatny Gabinet Lekarski i Wizyty Lekarskie Jan Ruxer, Lodz, Lódzkie
  - Synexus Polska Sp. z o.o., Katowice
  - Synexus Polska Sp. z. o.o., Lodz
  - SP ZOZ Centralny Szpital Kliniczny UM w Lodzi, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Synexus Polska Sp. z o.o., Poznan
  - Synexus Polska Sp. z o.o., Warsaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw
- Serbia (7):
  - Clinical Hospital Centre Zemun, Zemun, Belgrade
  - Clinical Centre Nis, Niš, Nišavski Okrug
  - Clinical Center Vojvodina, Novi Sad, Vojvodina
  - Military Medical Academy, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - MSB General hospital - Clinical Research Center, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- South Africa (5):
  - Iatros International, Bloemfontein, Free State
  - Charlotte Maxeke Johannesburg Hospital, Soweto, Gauteng
  - Office of Gulam Hoosain Vally, Durban, KwaZulu-Natal
  - Tiervlei Trial Centre, Bellville, Cape Town, Western Cape
  - Dr J.M. Engelbrecht Trial Site, Somerset West, Western Cape
- South Korea (6):
  - Chungnam National University Hospital - Nephrology, Daejeon, Daejeon Gwang'yeogsi [Taejon-Kwangyokshi]
  - National Health Insurance Service Ilsan Hospital - Nephrology, Goyang-si, Gyeonggido [Kyonggi-do]
  - Seoul National University Hospital - Nephrology, Jongno-gu, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Gangnam Severance Hospital, Yonsei University Health System - Internal Medicine, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Samsung Medical Center - Nephrology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
- Spain (10):
  - Hospital público da Mariña, Burela de Cabo, Lugo
  - Hospital Ribera Polusa, Burela de Cabo, Lugo
  - Consorcio Hospital General Universitario de Valencia, Valencia, Valenciana, Comunidad
  - FUNDACION PUIGVERT - Nephrology Department, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Y Politécnico La Fe, Valencia
- Taiwan (5):
  - Taichung Veterans General Hospital - Nephrology, Taichung, Taichung Municipality
  - National Taiwan University Hospital - Nephrology, Taipei, Taipei Special Muncipality
  - China Medical University Hospital - Nephrology - Taichung, Taichung
  - Taipei Medical University - Shuang Ho Hospital - Nephrology, Taipei
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Nephrology, Taoyuan District

IPD SHARING:
Plan to Share IPD: No